CLINICAL TRIAL: NCT04535739
Title: A Prospective Randomized Controlled Study for Prophylactic Cranial Irradiation After Chemotherapy and Thoracic Radiation Therapy in Patients With Extensive-stage Small Cell Lung Cancer
Brief Title: PCI for Patients With ES-SCLC After RCT:a Prospective Randomized Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zongmei Zhou, clinical professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-184/1440
Record Dates: First submitted 2020-08-28; First posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2019-10

CONDITIONS: Small-cell Lung Cancer
Keywords: small cell lung cancer; Brain Metastases
MeSH Terms: conditions — Small Cell Lung Carcinoma; Brain Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCI group (Experimental): patients received 4-6 circles of chemotherapy of EP or EC，and patients with complete remission or partial remission (more than 1 site) after chemotherapy，patients received thoracic radiotherapy and prophylactic cranial irradiation。
  Interventions: Radiation: prophylactic cranial irradiation
- control group (Other): patients received 4-6 circles of chemotherapy of EP or EC，and patients with complete remission or partial remission (more than 1 site) after chemotherapy，patients received thoracic radiotherapy。
  Interventions: Radiation: prophylactic cranial irradiation

INTERVENTIONS:
Radiation: prophylactic cranial irradiation — 25Gy/2.5Gy/10f were given for PCI patients

SUMMARY:
prophylactic cranial irradiation （PCI）was verified to decrease the brain metastases rates and improve the overall survival（OS）for patients with limited stage small cell lung cancer.We hypothesis that patients with extensive-stage small cell lung cancer after chemotherapy and thoracic radiation can also benefit from PCI.

DETAILED DESCRIPTION:
Patients with extensive-stage small cell lung cancer achieving CR or PR after chemotherapy and thoracic radiation therapy were randomly divided into observation group and prophylactic cranial irradiation (PCI) group to evaluate the effect of PCI on survival after radiation therapy for thoracic lesions. To preliminarily analyze the clinical characteristics of patients who would benefit from thoracic radiation therapy plus PCI. To explore the optimal treatment modality after chemotherapy + thoracic radiation therapy in patients with extensive-stage SCLC.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old,KPS≥70
* Pathological or cytological diagnosis of stage IV small cell lung cancer (by using AJCC 7th edition staging criteria);
* 1-3 extra-cranial metastatic organs before chemotherapy; 4-6 cycles of CE or EP ；
* CR or PR after chemotherapy；
* no grade ≥II side effects;
* the estimated overall survival time ≥ 3 months;
* no serious medical disease or major organ dysfunction.

Exclusion Criteria:

* Patients with brain or nervous system metastases;
* Presence of high grade radiation comorbidities;
* Patients who are pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 414 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
overall survival | 2 year
  rate of patients survival in 2 years

SECONDARY OUTCOMES:
progression-free survival | 2 year
  the rate of patients survival from the treatment to death or progress
brain metastases rates | 2 year
  Cumulative incidence of brain metastases over 2 year
side effect | 2 year
  HLVT

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China